CLINICAL TRIAL: NCT06253208
Title: Postoperative Analgesia in Laparoscopic Sleeve Gastrectomies: Laparoscopic Versus Ultrasound-guided Transversus Abdominis Plane Block
Brief Title: Laparoscopic Versus Ultrasound Guided Block in Sleeve Gastrectomy
Status: Recruiting | Type: Observational
Sponsor: Biruni University (Other)
Responsible Party: Principal Investigator, ilke dolğun, anesthesia and reanimation, Biruni University
Other Study IDs: istinye
Record Dates: First submitted 2024-02-02; First posted 2024-02-12 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Postoperative Pain
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- laparoscopic block: laparoscopic transversus abdominis plane block
  Interventions: Procedure: postoperative pain
- ultrasound guided block: ultrasound guided transversus abdominis plane block
  Interventions: Procedure: postoperative pain

INTERVENTIONS:
Procedure: postoperative pain — Postoperative analgesia in laparoscopic sleeve gastrectomies: laparoscopic versus ultrasound-guided transversus abdominis plane block

SUMMARY:
Comparison of pain conditions in the first 24 hours after surgery in terms of two different analgesia methods

DETAILED DESCRIPTION:
Introduction and purpose:

Morbid obesity (MO) is a disease that has become a worldwide epidemic, and in the last three decades, the average body mass index (BMI) has increased by 0.4 kg/m2 per decade worldwide. Parallel to this situation, the number of obesity surgery operations is increasing steadily. In 2017, this number reached 228,000 surgeries in the United States. In particular, due to its technical simplicity and positive outcomes, laparoscopic sleeve gastrectomy (LSG) has become the dominant bariatric operation, accounting for approximately 60% of all bariatric procedures (1) These individuals are at high risk for postoperative adverse respiratory events, nosocomial infections, cardiovascular complications, and pulmonary embolism (the second leading cause of death in the bariatric surgery population). Therefore, given the increasing number of patients living with obesity and seeking elective weight loss surgery, it is crucial to understand and optimize the analgesic requirements of this patient population. However, no ideal analgesic regimen exists for this patient population and limited evidence-based recommendations (2) Pain management of the MO patient is an evolving issue and remains extremely important in terms of patient safety and possible addiction risk. Effective postoperative pain management is crucial to encouraging early walking and deep breathing, which are known to reduce the risk of complications. Multimodal analgesia has been advocated by many authors as part of Enhanced Recovery After Surgery (ERAS) programs to reduce the incidence and severity of postoperative pain (3).

Similar to the increase in the number of MOs over the past three decades, opioid use has also increased dramatically. In the United States, opioid overdose has become the leading cause of unintentional death, surpassing motor vehicle crashes. Frequently, the first exposure to opioids may occur during the perioperative period of an elective surgery. It has been reported that approximately 6-8% of opioid-naïve patients undergoing non-cancer procedures develop new persistent opioid use (1). Increased opiate use is associated with increased rates of delirium, ileus, urinary retention, and respiratory depression and may have strong addictive potential. Opioid-induced cardiopulmonary arrest usually occurs within the first 24 hours of surgery (3). Therefore, the surgical team has a critical role in patient management in terms of opioid-independent analgesia control.

To optimize pain control, multimodal anesthesia and regional analgesia have become key components of improved clinical recovery pathways and therefore recommended methods for perioperative pain control. One of these is the transversus abdominis plane (TAP) block, whose effectiveness has been proven in this patient group.

TAP blocks are widely used for intraoperative and postoperative analgesia in various abdominal and gynecological surgeries. There is evidence in the literature that TAP blocks are beneficial in laparoscopic (minimally invasive) surgeries such as laparoscopic cholecystectomy, hernia repair and laparoscopic colorectal resection (4-8). Similarly, in two of the studies demonstrating the feasibility of TAP blocks in laparoscopic bariatric surgery (9,10), it was shown that there was a decrease in pain scores and in another (9) it was shown that it reduced opioid consumption.

Traditionally, the TAP block is completed by an anesthesiologist at the beginning or end of surgery, using ultrasound guidance to improve the accuracy of visualization of the target anatomy and the spread of local anesthesia within the application area (US-TAP). However, in recent years, a new technique has been developed and started to be used during laparoscopic surgery, in which the surgeon can perform the TAP block under direct visualization: laparoscopy-guided TAP block (L-TAP). Numerous studies and technical reports describe this laparoscopic-assisted technique. Studies have shown that laparoscopic-assisted TAP blocks result in similar pain scores and postoperative opioid consumption but lead to shorter block performance time compared to ultrasound-guided block (11). Additionally, a statistically significant decrease was observed in the pain scores and opioid consumption of patients receiving laparoscopic-assisted TAP block compared to controls (12,13). Similarly, in a meta-analysis, it was stated that L-TAP provided comparable analgesia to US-TAP, and there was no statistically significant difference in pain scores at different times and during both rest and movement (14). According to the same meta-analysis, patients in most studies achieved adequate pain control, and 24-hour opioid consumption, incidence of postoperative nausea and vomiting, functional recovery, bowel function, and hospital stay rates did not differ significantly between the 2 methods.

ELIGIBILITY:
Inclusion Criteria:

* Patients who can tolerate general anesthesia and pneumoperitoneum.
* Patients who can give informed consent for surgery.
* Patients over 18 years of age
* patients with body mass index (BMI) > 30 kg/m2
* Patients with American Society of Anesthesiologists (ASA) physical status I and II

Exclusion Criteria:

* Patients allergic to local anesthetics.
* Patients with serious underlying cardiovascular disease (e.g. congestive heart failure, conduction disorders and ischemic heart disease).
* Patients with chronic kidney disease stage 3 or greater (creatinine clearance less than 60 mL/min).
* Patients who have had previous abdominal surgery, including resection of the esophagus, stomach, liver and pancreas.
* Patients with chronic pain and chronic opioid use
* Patients with ASA class IV
* patients with psychiatric disorders
* pregnant or breastfeeding patients
* patients with a history of seizures

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 50 patients over the age of 18 who will undergo laparoscopic sleeve gastrectomy will be included in the study.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-01-01 (Actual); Primary Completion 2024-04-24 (Estimated); Study Completion 2024-06-24 (Estimated)

PRIMARY OUTCOMES:
postoperative pain | 4 month
  postoperative pain

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Okut G, Turgut E, Kaplan K, Bag YM, Akbas S, Sumer F, Kayaalp C. Does laparoscopic-guided transversus abdominis plane block have an effect on postoperative pain and recovery after sleeve gastrectomy? Eur Rev Med Pharmacol Sci. 2022 Aug;26(15):5406-5412. doi: 10.26355/eurrev_202208_29408. PMID 35993635
- [Result] Hamid HK, Emile SH, Saber AA, Ruiz-Tovar J, Minas V, Cataldo TE. Laparoscopic-Guided Transversus Abdominis Plane Block for Postoperative Pain Management in Minimally Invasive Surgery: Systematic Review and Meta-Analysis. J Am Coll Surg. 2020 Sep;231(3):376-386.e15. doi: 10.1016/j.jamcollsurg.2020.05.020. Epub 2020 Jun 2. PMID 32502615
- [Result] Venkatraman R, Saravanan R, Dhas M, Pushparani A. Comparison of laparoscopy-guided with ultrasound-guided subcostal transversus abdominis plane block in laparoscopic cholecystectomy - A prospective, randomised study. Indian J Anaesth. 2020 Dec;64(12):1012-1017. doi: 10.4103/ija.IJA_528_20. Epub 2020 Dec 12. PMID 33542563